CLINICAL TRIAL: NCT00689806
Title: Evaluation of Lovastatin in Severe Persistent Asthma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study never opened
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15427A; UL1RR024999 (NIH)
Record Dates: First submitted 2008-05-23; First posted 2008-06-04 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Severe Persistent Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Lovastin (Active Comparator)
  Interventions: Drug: Lovastatin

INTERVENTIONS:
Drug: Lovastatin — Lovastatin 20 mg extended release (or placebo) by mouth once daily for weeks 1-4. Liver function test will be checked at week 4 follow up visit. If LFTs are not > 3 times the upper limit of normal, then the subject will have the dose of extended release lovastatin increased to 60 mg once a day for weeks 4-12
  Arms: Lovastin
Drug: Placebo — Placebo by mouth once daily for weeks 1-4.
  Arms: Placebo

SUMMARY:
This study has two purposes:

1. to determine whether lovastatin, a commonly used medication to lower cholesterol in the blood, can produce beneficial changes in airway inflammation and in the airway smooth muscle
2. to examine whether lovastatin will have favorable changes in asthma symptoms of patients with moderate or severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years to <65 years
* Severe persistent asthma (per 2002 National Asthma Education and Prevention Program guidelines)
* Treatment with daily fluticasone (500 ug BID) and salmeterol (50 ug BID) during the past 4 or more weeks
* Pre-bronchodilator FEV1 <80% predicted
* Post-bronchodilator improvement in FEV1 of at least 12% and 200 mL or a PC20 to methacholine of <8 mg/mL
* Evidence of inadequate asthma control in the past 2 weeks: use of rescue inhaler > 4 days and >8 occasions in the past 2 weeks, daytime asthma symptoms > 4 days in the past 2 weeks, or 1 or more nocturnal awakening in the past 2 weeks
* No evidence of alternate diagnosis (e.g., sarcoidosis, eosinophilic pneumonia) on bronchoscopy performed as part of routine care in the Refractory Obstructive Lung Disorders clinic.
* Completed research bronchoscopy while on current dose of daily fluticasone and salmeterol within 4 weeks of meeting other inclusion criteria. Note: many patients in the ROLD clinic require a bronchoscopy to confirm the diagnosis of asthma and exclude other diagnosis (e.g., sarcoidosis). These patients are asked to participate in a research protocol (separate from this proposal) that allows investigators to collect additional samples (endobronchial biopsies, bronchoalveolar lavage fluid, endobronchial brushings) at the end of the clinical portion of the bronchoscopy {IRB protocol # 15361A entitled, "Airway inflammation in refractory obstructive lung disease (ROLD): understanding markers of inflammation and remodeling"}. This protocol was recently submitted to the IRB in March 2007.

Exclusion Criteria:

* Pregnancy or lactation
* Severe metabolic disease
* Other respiratory or inflammatory disorders (sarcoidosis, emphysema)
* Hypokalemia, dehydration
* Uncontrolled seizure disorder ( 2 or more seizures in last year)
* Major surgery, trauma
* Pre-existing liver disease (AST or ALT >10% above the upper limit of normal)
* Elevated CK (>50% above the upper limit of normal)
* History of alcohol abuse
* Current smokers or ex-smokers with > 10 pack-years of smoking
* Partial ileal bypass surgery
* Concurrent treatment with drugs known to be have potential interactions or associated with rhabdomyolysis (Cimetadine, danazole, delavaridine, diltiazem, fenofiibrate, nefazodone, niacin, protease inhibitors, quinipristoline/dalfopristin, ranolazine, rifampin, telbivudine, telithromycin)
* HIV patients taking protease inhibitors
* History of allergy or intolerance to statin
* Use of 1 or more doses of any cholesterol lowering medication in the previous 12 weeks
* Clinical indication for treatment with statins

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Changes in airway smooth muscle biology and inflammatory measures | 12 Weeks

SECONDARY OUTCOMES:
Changes in asthma control, lung function and quality of life from the baseline visit to the end of the follow-up period | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Camoretti-Mercado, Ph.D., Principal Investigator — University of Chicago